CLINICAL TRIAL: NCT02616796
Title: Effects of Social Gaze Training on Brain and Behavior in Fragile X Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Scott Hall, Associate Professor, Stanford University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 31648
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Fragile X Syndrome; Intellectual Disability
MeSH Terms: conditions — Fragile X Syndrome; Intellectual Disability

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social gaze training (Experimental): Appropriate social gaze behavior will be reinforced using the principles of Applied Behavior Analysis.
  Interventions: Behavioral: Social gaze training
- No Training (No Intervention): Appropriate social gaze behavior will not be reinforced.

INTERVENTIONS:
Behavioral: Social gaze training — Appropriate social gaze behavior will be shaped using the principles of Applied Behavior Analysis.
  Arms: Social gaze training

SUMMARY:
The purpose of the study is to evaluate a 2-3 day treatment probe targeted to improving social gaze behavior in children with fragile X syndrome (FXS). The investigators will use the principles of Applied Behavior Analysis (ABA) to shape appropriate social skills. Importantly, the investigators propose to examine the effects of this treatment probe on brain and behavior.

ELIGIBILITY:
Inclusion Criteria:

1. Boys diagnosed with fragile X syndrome
2. Boys with intellectual disability who do not have FXS or other known genetic disorder associated with intellectual disability
3. Age 8 to 18 years inclusive
4. Ability to travel to Stanford
5. Vineland Adaptive Behavior Scales standard score between 50 and 75 points

Exclusion Criteria:

1. Sensory impairments, or any other serious medical or neurological condition that affects growth or development (e.g., seizure disorder, diabetes, congenital heart disease).
2. Materials in body that would preclude an MRI scan (e.g., dental braces).

Ages: 8 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2015-04; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Percentage of social gaze aversion recorded during the social challenge | 3 days
Heart rate recorded during the social challenge | 3 days
Total t-score on the Social Responsiveness Scale (SRS) | 4 weeks

SECONDARY OUTCOMES:
Verbal responses and pauses in conversation observed during the social challenge | 3 days
Fractional Amplitude of Low Frequency fluctuations (fALLF) measured in the insular cortex | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Gannon CE, Britton TC, Wilkinson EH, Hall SS. Improving social gaze behavior in fragile X syndrome using a behavioral skills training approach: a proof of concept study. J Neurodev Disord. 2018 Aug 28;10(1):25. doi: 10.1186/s11689-018-9243-z. PMID 30153790